CLINICAL TRIAL: NCT00985868
Title: A CCLG/Cancer Research UK Phase I Trial of AT9283 (a Selective Inhibitor of Aurora Kinases) Given for 72 Hours Every 21 Days Via Intravenous Infusion in Children and Adolescents With Relapsed and Refractory Solid Tumors
Brief Title: AT9283 in Children and Adolescents With Relapsed and Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000653387; UKM-ICRF-CR0708-11; CRUK-CR0708-11; EUDRACT-2008-005542-23; EU-20980
Record Dates: First submitted 2009-09-26; First posted 2009-09-29 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

INTERVENTIONS:
Drug: multikinase inhibitor AT9283
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: AT9283 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of AT9283 in children and adolescents with relapsed and refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and tolerability of Aurora kinase inhibitor AT9283 by characterizing the dose-limiting toxicities in children and adolescents with relapsed and refractory solid tumors.
* To determine the maximum-tolerated dose of this regimen in these patients.

Secondary

* To determine the pharmacokinetic parameters of this regimen in these patients.
* To demonstrate the pharmacodynamic (PD) activity of this regimen in these patients by studying its effects in surrogate tissue.
* To assess preliminary evidence of activity of this regimen by using appropriate objective tumor measurements in these patients.

Tertiary

* To demonstrate the PD activity of this regimen in these patients by studying its effects in both surrogate and tumor tissue (skin punch, bone marrow, and tumor biopsies).

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive Aurora kinase inhibitor AT9283 IV over 72 hours on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.If a patient is benefiting from treatment with AT9283 (i.e. has stable or responding disease as measured by RECIST) and the benefit risk balance is considered acceptable then further treatment may be given.

Blood and skin tissue samples are collected at baseline and periodically during treatment for pharmacokinetic studies and pharmacodynamic and biomarker (M30, M65, pHH53, p53, PCNA and Ki67) analysis by IHC and ELISA assays.

After completion of study therapy, patients are followed up periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor meeting 1 of the following criteria:

  * Refractory to conventional treatment
  * Disease for which no conventional therapy exists
* Patients with CNS tumors must be on a stable or decreasing dose of dexamethasone for ≥ 1 week before study entry

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 OR Lansky Play PS 70-100% (> 50% is acceptable if it is due to a stable neurological deficit or CNS tumor)
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Serum bilirubin < 1.5 times upper limit of normal (ULN)
* Creatinine kinase normal
* ALT or AST < 2.5 times ULN (≤ 5 times ULN if due to tumor)
* Creatinine clearance/EDTA-measured GFR ≥ 60 mL/min
* Sufficient blood volume to undergo the blood-sampling regimen specified by the protocol that, in the opinion of the investigator, will not jeopardize patient's safety
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 4 weeks before, during, and for 6 months after completion of study therapy
* Not at high medical risk because of non-malignant systemic disease, including active uncontrolled infection
* Not known to be serologically positive for hepatitis B or C or HIV
* Fractional shortening of > 29% on echocardiogram
* LVEF ≥ 50%
* No history of allergy or auto-immune disease
* No congenital heart disease
* No other condition that, in the investigator's opinion, would not make the patient a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 4 weeks since prior radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, or chemotherapy (6 weeks for investigational medicinal products, 2 weeks for vincristine)
* More than 3 months since prior autologous stem cell transplantation
* No prior allogenic bone marrow transplantation
* No prior extensive radiotherapy to > 25% of bone marrow
* No prior Aurora kinase inhibitor
* No prior major thoracic or abdominal surgery from which the patient has not yet recovered
* No prior or concurrent participation in another interventional clinical trial

  * Participation in an observational study allowed
* No other concurrent anticancer therapy or investigational drugs

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2016-01-25 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities
Maximum-tolerated dose

SECONDARY OUTCOMES:
Pharmacokinetic parameters and the correlation between them and toxicity and/or efficacy
The magnitude and duration of biomarkers (M30 and M65 ELISA) change after AT9283 administration
Objective tumor response according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Darren Hargrave, MD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham, England
  - Leeds General Infirmary, Leeds, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Great North Children's Hospital, Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Royal Marsden - Surrey, Sutton, England